CLINICAL TRIAL: NCT07015151
Title: Lyon Initiative for the Mobile Demedicalized Initiation of Lung Cancer Screening
Brief Title: Mobile Lung Cancer Screening
Acronym: MobILYAD
Status: Recruiting | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL22_0467; 2025-A00673-46 (Other: ID-RCB)
Record Dates: First submitted 2025-06-03; First posted 2025-06-11 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-09

CONDITIONS: Lung Cancer Prevention
Keywords: Prevention; Lung cancer; screening; tobacco
MeSH Terms: conditions — Lung Neoplasms | interventions — Spirometry

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — The following types of biospecimens will be retained for ancillary analyses:
  * Exhaled breath condensate
  * Blood samples
  These specimens will be collected at baseline and at the end of the intervention phase, then stored for subsequent analysis in the context of the Bio-ILYAD study (biobank).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Mobile Screening Group: Participants receiving lung cancer screening via a mobile unit (truck) operated by trained nurses. This includes spirometry, blood pressure measurement, blood cholesterol testing, low-dose CT scan, and optional biospecimen collection.
  Interventions: Diagnostic Test: Low-dose Chest CT Screening; Diagnostic Test: Spirometry; Diagnostic Test: Cardiovascular Risk Assessment; Behavioral: Smoking Cessation Support; Other: Optional Biospecimen Collection (Bio-ILYAD)
- Non-Mobile Screening Group: Participants receiving the same screening procedures at a fixed hospital-based site (Lyon Sud), with possible involvement of medical or non-medical staff depending on availability.
  Interventions: Diagnostic Test: Low-dose Chest CT Screening; Diagnostic Test: Spirometry; Diagnostic Test: Cardiovascular Risk Assessment; Behavioral: Smoking Cessation Support; Other: Optional Biospecimen Collection (Bio-ILYAD)

INTERVENTIONS:
Diagnostic Test: Low-dose Chest CT Screening — Participants undergo a low-dose chest CT scan to screen for early lung cancer and assess associated conditions (emphysema, coronary calcifications, osteoporosis).
Diagnostic Test: Spirometry — Assessment of lung function through spirometry, with optional plethysmography and diffusion testing to detect COPD and PRISM patterns.
Diagnostic Test: Cardiovascular Risk Assessment — Cardiovascular risk is evaluated using SCORE2/SCORE2-OP tools, based on blood pressure and cholesterol levels.
Behavioral: Smoking Cessation Support — Active smokers receive a structured smoking cessation intervention, including a baseline consultation and up to two follow-up sessions (which may be remote).
Other: Optional Biospecimen Collection (Bio-ILYAD) — Optional collection of blood and exhaled breath condensate for future analysis of biomarkers in lung cancer detection.

SUMMARY:
Lung cancer screening using low-dose CT (LDCT) has been shown to reduce mortality in high-risk populations. In 2022, the French National Cancer Institute (INCa) issued guidelines recommending screening for individuals aged 50-74 with a history of heavy smoking, including current smokers or those who quit less than 15 years ago. A national pilot program (IMPULSION) will be launched in 2025.

Lung cancer incidence is strongly correlated with socioeconomic status, yet underserved populations remain difficult to engage in screening programs. Mobile health units using a "reach-out" strategy have demonstrated effectiveness in other countries (UK, Brazil, USA). In France, this approach has been used for breast cancer screening via mobile mammography units.

The MobILYAD project aims to compare two screening modalities- a mobile demedicalized unit (CT-equipped van with trained nurses) and a conventional hospital-based unit- to assess the effectiveness of mobile screening in reaching socially disadvantaged populations.

ELIGIBILITY:
Inclusion Criteria * :

* Persons aged over 50 and under 75 (74 years of age or older).
* Active smokers or former smokers who quit less than 15 years ago.
* Persons whose consumption is estimated at 20 packs/year or more, down to ≥15 cigarettes/day for a duration of consumption of ≥25 years and up to ≥10 cigarettes/day for ≥30 years, which takes into account the predominance of duration of consumption over quantity consumed in the risk of lung cancer. A pack-year corresponds to the consumption of one pack of 20 manufactured cigarettes per day for one year. A multiplier coefficient will be taken into account depending on the mode of consumption: Rolled cigarettes: 2; Cigarillos: 3; Cigars: 4; Pipes: 2.5; Hookahs: 25.
* Persons affiliated with social security. - Person having signed their consent to participate in the study after having received full information about it, including the risks associated with participation.

  * Exclusion Criteria * :
* Individuals with severe comorbidities contraindicating lung cancer investigations and/or treatment (including surgery or stereotactic radiotherapy);
* Individuals with impaired general condition (PS 2 and above);
* Individuals with dyspnea at rest (mMRC4);
* Individuals with a history of cancer undergoing active surveillance by chest computed tomography (CT or PET scan); personal history of lung cancer (lifetime);
* Individuals with symptoms suggestive of lung cancer (hemoptysis, unexplained weight loss, recent onset or change in respiratory symptoms, etc.);
* Individuals refusing to participate in the study
* Individuals withdrawing their consent.

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adults aged 50 to 74 years with a significant history of smoking, currently smoking or former smokers who quit within the past 15 years. The study targets individuals eligible for lung cancer screening per national guidelines, with a focus on those from socially deprived backgrounds. Recruitment will be carried out through a mobile screening unit or a fixed hospital site, depending on geographic location.
Sampling Method: Non-Probability Sample
Enrollment: 4312 (Estimated)
Dates: Start 2025-06-12 (Actual); Primary Completion 2028-09 (Estimated); Study Completion 2028-09 (Estimated)

PRIMARY OUTCOMES:
Proportion of socially deprived participants included in the mobile screening group | Baseline (Day 0)
  The percentage of participants with an EPICES score ≥ 4 (indicating social vulnerability) in the mobile screening arm, compared to the non-mobile arm.

SECONDARY OUTCOMES:
Participation by socio-demographic profile | Inclusion
  Comparison of participants' characteristics between the two modalities (smoking status, age, sex, socio-professional category, income level, education, perceived ethnic identity, geographic isolation, presence of a general practitioner).
Mobile feasibility | Throughout inclusion period
  Feasibility of the mobile screening pathway, assessed by the attendance rate (proportion of invited participants who attend the mobile unit) and the completion rate (proportion of those attendees who complete the full screening process). Both will be reported separately as percentages.
  Unit of Measure: Percentage of participants (%)
Feasibility of task-shifting to nurses | Throughout inclusion period
  Rate of recourse to a physician and participant satisfaction in each modality.
Adherence to intermediate CT scans | Month 1, Month 3, Month 6 if clinically indicated
  Proportion of participants who undergo intermediate follow-up CTs when required.
Adherence to 12-month CT scan | At Month 12
  Proportion of participants who complete the scheduled CT scan at one year.
Adherence to tobacco cessation consultations | Over 12 months
  Proportion of active smokers who attend the initial and, if applicable, follow-up cessation visits.
Smoking cessation success | At 12 months
  Self-reported complete tobacco cessation at 12 months.
Rate of positive screening | Up to 3 months post-initial CT
  Proportion of participants with positive CT findings and subsequent medical workup.
Lung cancer incidence | Over 12 months
  Number and percentage of participants diagnosed with lung cancer during the 12-month follow-up.
COPD detection relevance | Baseline and 12 months
  Rate of new COPD diagnoses and associated therapeutic modifications; respiratory morbidity and mortality over 12 months.
Cardiovascular risk detection relevance | Baseline and 12 months
  Rate of high-risk participants identified, therapeutic implications, cardiovascular events over follow-up.
Creation of biobank (Bio-ILYAD) | At inclusion
  Proportion of participants consenting to blood and exhaled air sample collection for future biomarker research.
Lung cancer staging | Within 12 months
  Distribution of lung cancer cases by stage at diagnosis (I-IV), as recorded in clinical reports. Number of participants per stage
Histological type of diagnosed lung cancers | Within 12 month
  Categorization of diagnosed lung cancers by histological type (e.g., adenocarcinoma, squamous cell carcinoma, small cell). Number of participants per histological category
Initial treatment of diagnosed lung cancers | Within 3 months of diagnosis
  Description and frequency of initial treatment modalities (e.g., surgery, radiotherapy, systemic therapy). Number of participants per treatment type

OTHER OUTCOMES:
Creation of CT image database | Baseline, 6 months and 12 months
  Establishment of a thoracic imaging repository for AI model training and teaching purposes.

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - " Centre de dépistage mobile " - Hôpital Lyon Sud, Pierre-Bénite
  - Service de Pneumologie " Centre de dépistage non mobile " - Hôpital Lyon Sud, Pierre-Bénite

IPD SHARING:
Plan to Share IPD: Undecided
A decision on sharing individual participant data has not yet been made. Data sharing will depend on sponsor policy, ethical approval, and compliance with applicable regulations.